CLINICAL TRIAL: NCT01414946
Title: THE PROTEIN SPARING EFFECT OF PERIOPERATIVE NUTRITION: How Important is the Patient's Catabolic State Before Surgery and do we Need Glucose?
Brief Title: The Effect of Intravenous Nutrition in Patients Undergoing Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Thomas Schricker, Department of Anaesthesia, Royal Victoria Hospital, MUHC
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIHR-2011
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Postoperative Protein Catabolism
MeSH Terms: interventions — Glucose; Amino Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose and amino acids (Experimental): Perioperative nutrition with glucose and amino acids
  Interventions: Other: Intravenous nutrition with glucose and amino acids
- Amino acids only (Active Comparator): Perioperative nutrition with amino acids only
  Interventions: Other: Intravenous nutrition with amino acids

INTERVENTIONS:
Other: Intravenous nutrition with glucose and amino acids — Glucose and amino acids intravenously starting 20 hours before the operation until the second postoperative day. Glucose provides 50% and amino acids 20% of each patient's measured resting energy expenditure.
  Arms: Glucose and amino acids
Other: Intravenous nutrition with amino acids — Amino acids intravenously starting 20 hours before the operation until the second postoperative day. Amino acids providing 20% of each patient's measured resting energy expenditure.
  Arms: Amino acids only

SUMMARY:
Loss of muscle protein and mass are the main causes of fatigue after bowel surgery which may result in a longer hospital stay and a higher rate of complications. This problem is especially important for patients after surgery for bowel cancer because cancer itself causes a waste of muscle protein. Anesthesiologists can decrease these negative effects of surgery by choosing the type of pain treatment (analgesia) and by giving nutrition (sugar and protein). Our group recently observed that optimal pain relief with epidural catheters (these are placed in the so called epidural space, which lies between the spine and the skin of the back) in combination with a low calorie protein diet intravenously (through the vein) maintains the body's protein stores after bowel surgery.

The goal of our new research program is to find out whether this protein saving effect depends on how protein depleted the patient is before surgery. In other words we would like to answer the question: do cancer patients who show protein wasting before the operation benefit more from feeding than patients who show no signs of protein wasting? A second goal of this program is to find out if we need to use sugar as part of the diet or whether the infusion of protein alone is sufficient. Just giving protein would make feeding not only easier but also would avoid the increase in the patient's own blood sugar during and after the operation, which typically occurs when sugar is given intravenously during that period.

DETAILED DESCRIPTION:
1. Goals The overall goal of perioperative nutrition support is to abolish protein wasting and to promote anabolic processes by directing amino acids into protein synthesis rather than oxidation. Protein repletion and enhancement of anabolism appear to be particularly important in cancer patients who enter major abdominal surgery in a catabolic state.
2. Objectives The objectives of this research program are

   * to examine whether the anabolic effects of hypocaloric nutrition depend on the degree of catabolism before the operation and thus identify patients who benefit the most from perioperative nutrition support (study I)
   * to investigate whether excluding glucose from hypocaloric nutrition, i.e. infusing an isonitrogenous amount of amino acids without glucose avoids hyperglycemia and, thus, accentuates the patient's anabolic response to feeding (study II).

In order to confirm the validity of our assumptions we will perform two consecutive studies in two distinct patient populations. For the assessment of the patients' catabolic state and obtaining insight into the biochemical mechanisms, whereby the effects of nutrition are mediated, stable isotope tracer kinetics will be applied. Using primed continuous infusions of L-[1-13C]leucine and [6,6-2H2]glucose we will quantitate the whole body dynamics of protein and glucose metabolism, i.e. protein breakdown, amino acid oxidation, protein synthesis, glucose production and glucose uptake before and after surgery. A positive protein balance (difference between protein synthesis and protein breakdown) will be used as an indicator of anabolism. Anabolic processes at the organ level (liver, muscle), i.e. fractional synthesis rates of the acute phase proteins albumin and fibrinogen and muscle protein synthesis will be determined using L-[2H5]phenylalanine infusions. Skeletal muscle protein catabolism will be characterized by measuring the mRNA expression of ubiquitin and two of its key ligases in muscle (MAFbx/atrogen-1 and MuRF-1).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists <3
* colorectal surgery for non-metastatic colorectal carcinoma including right and left hemicolectomy, transverse, subtotal and total colectomy, sigmoid resection
* ability to give informed consent

Exclusion Criteria:

* signs of severe malnutrition or obesity: body mass index <18 or >25 >10% involuntary body weight loss over the preceding 6 months serum albumin <21 g/L
* significant cardiorespiratory, hepatic, renal and neurological disease
* ingestion of drugs known to affect protein, glucose and lipid metabolism (for example steroids)
* musculoskeletal or neuromuscular disease
* severe anemia (hemoglobin <10 g/dL)
* pregnancy
* history of severe sciatica or back surgery or other conditions which
* contraindicate the use of epidural catheters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
protein balance | two days after surgery

SECONDARY OUTCOMES:
albumin synthesis | two days after surgery
fibrinogen synthesis | two days after surgery
total plasma protein synthesis | two days after surgery
mRNA expression of ubiquitin | two days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schricker, MD PhD, Principal Investigator — Department of Anaesthesia, McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Schricker T, Wykes L, Meterissian S, Hatzakorzian R, Eberhart L, Carvalho G, Meguerditchian A, Nitschmann E, Lattermann R. The anabolic effect of perioperative nutrition depends on the patient's catabolic state before surgery. Ann Surg. 2013 Jan;257(1):155-9. doi: 10.1097/SLA.0b013e31825ffc1f. PMID 22878551